CLINICAL TRIAL: NCT07098546
Title: Diagnostic Value of Right Ventricular 'Bubble Time' in Pulmonary Embolism
Brief Title: 'Bubble Time' in Pulmonary Embolism
Status: Active, not recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Marmara University Pendik Training and Research Hospital (Other); Gazi University (Other); Akdeniz University Hospital (Other)
Responsible Party: Principal Investigator, Mümin Murat Yazıcı, Emergency Specialist, Principal Investigator, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: Mumin Murat YAZICI
Record Dates: First submitted 2025-07-04; First posted 2025-08-01 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Tanısal değerlilik
Keywords: pulmonary embolism; bubble time; pocus
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will be multi-centre and prospectively planned. All patients who undergo contrast-enhanced computed tomography in the emergency department with a preliminary diagnosis of pulmonary embolism and who do not meet the exclusion criteria will be included in the study. Informed consent will be obtained from all patients prior to the study. Patients included in the study will undergo bedside ultrasound to assess bubble time, right ventricle-left ventricle ratio, presence of a septal defect, and tricuspid insufficiency, and the diagnostic value of these findings will be evaluated. The bedside ultrasound will be part of the emergency department critical care examination, will not incur any costs for the institution, and will be performed and evaluated by an emergency medicine specialist and assistant.

DETAILED DESCRIPTION:
The study will be multi-centre and prospectively planned. All patients who undergo contrast-enhanced computed tomography in the emergency department with a preliminary diagnosis of pulmonary embolism and who do not meet the exclusion criteria will be included in the study. Informed consent will be obtained from all patients prior to the study. Patients included in the study will undergo bedside ultrasound to assess bubble time, right ventricle-left ventricle ratio, presence of a septal defect, and tricuspid insufficiency, and the diagnostic value of these findings will be evaluated. The bedside ultrasound will be part of the emergency department critical care examination, will not incur any costs for the institution, and will be performed and evaluated by an emergency medicine specialist and assistant.

ELIGIBILITY:
Inclusion Criteria:

- All patients presenting to the emergency department with any symptoms, undergoing pulmonary CT angiography due to suspected pulmonary embolism or evaluated as having a strong likelihood of embolism when CT cannot be performed will be included in the study.

Exclusion Criteria:

* Patients under the age of 18
* Patients with a severe history of tricuspid insufficiency
* Patients with a severe of pulmonary hypertension
* Patients with a severe of right heart failure
* Patients without an echocardiographic report approved by cardiology within 48 hours after emergency admission
* Patients in whom ultrasonographic measurements cannot be performed
* Patients who refuse diagnosis and treatment voluntarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1.000.000
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Bubble time | through study completion, an average of six months
  The diagnostic value of bubble time
bubble time in pulmonary embolism | through study completion, an average of six months
  The diagnostic value of bubble time in pulmonary embolism

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan Üniversitesi Rize Eğitim ve Araştırma Hastanesi, Rize, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen A, Li T, Bielawa N, Nello A, Gold A, Gorlin M, Nelson M, Carlin E, Rolston D. Right Ventricular "Bubble Time" to Identify Patients With Right Ventricular Dysfunction. Ann Emerg Med. 2024 Aug;84(2):182-194. doi: 10.1016/j.annemergmed.2024.02.005. Epub 2024 Apr 10. PMID 38597847